CLINICAL TRIAL: NCT02939677
Title: Can Targeted Exercise Improve Knee Strength in Patients With Persisting Hamstring Deficiency Following ACL-reconstruction? - A Randomized Controlled Trial
Brief Title: Can Targeted Exercise Improve Knee Strength Following ACLR (RATE)
Acronym: RATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Bo Bregenhof, M.D. Cand. Med. Ph.D student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SDUSF-2014-5 - (10); SDUSF-2015-20 - (115) (Other: PhD School - Faculty of Health Sciences, SDU)
Record Dates: First submitted 2016-10-04; First posted 2016-10-20 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Rupture of Anterior Cruciate Ligament; Muscle Degeneration; Gait, Unsteady
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted exercise (Other): Targeted exercise intervention
  Interventions: Other: Targeted exercise
- care as usual (No Intervention): home based exercises

INTERVENTIONS:
Other: Targeted exercise — 12 weeks of targeted and supervised exercise intervention vs. "care as usual" (home based exercises)
  Arms: Targeted exercise

SUMMARY:
Anterior cruciate ligament reconstruction (ACLR) is high volume surgery, carried out in about 2800 patients annually in Denmark per year. ACLR patients (using hamstring auto-graft) have persistent hamstring strength deficiency when evaluated more than 1-2 years after ACL-reconstruction. The investigators have designed this randomized controlled trial (RCT) with the main purpose to investigate the effect of a targeted muscle strength exercise intervention on the neuromuscular rehabilitation of ACLR-patients compared with 'care-as- usual'.

The study is designed as a prospective, superiority, parallel-group with balanced randomization (1:1) RCT (Level of evidence: II) with blinded allocation, and outcome assessment according to the CONSORT statement (Consolidated Standards of Reporting Trials). 50 patients with ACL reconstruction and persistent hamstring muscle deficiency, will be recruited at the outpatient clinic 1-year follow-up, and allocated to one of two 12 weeks' interventions, either a) the supervised progressive strength and neuromuscular exercise group (SNG) with supervised training twice weekly. Or b) the control group (CON) receiving patient education based on a home-based exercise regime of low intensity, defined as 'care as usual'. Outcome measures include, maximal isometric knee flexor muscle strength (primary outcome), knee extensor strength, and the Knee injury and Osteoarthritis Outcome Score (KOOS) (secondary outcomes). In addition, the following explorative outcomes will be investigated; hamstring to quadriceps strength ratios, the International Knee Documentation Committee Subjective Knee Form (IKDC), magnetic resonance imaging (MRI) to evaluate tendon regeneration of the hamstrings and finally kinetic/kinematic biomechanical outcomes of knee related functional tasks.

To the investigators knowledge, this is the first RCT to investigate the efficacy of combined progressive resistance training and neuromuscular exercise in the late rehabilitation phase in patients demonstrating persistent limb-to-limb knee muscle asymmetry following ACLR. Reduced hamstring strength represents a potential risk factor for secondary ligament rupture and accelerated progression of osteoarthritis (OA). If deemed effective, the intervention paradigm introduced in this study may help to improve current treatment strategies.

DETAILED DESCRIPTION:
Detailed study description available in the published study protocol:

"The effect of targeted exercise on kneemuscle function in patients with persistent hamstring deficiency following ACL reconstruction - study protocol for a randomized controlled trial".

Bo Bregenhof1,3* , Uffe Jørgensen1, Per Aagaard2, Nis Nissen3, Mark W. Creaby4, Jonas Bloch Thorlund2, Carsten Jensen3, Trine Torfing5 and Anders Holsgaard-Larsen1 Published: Trials. 2018; 19: 75. Published online 2018 Jan 26. doi: 10.1186/s13063-018-2448-3

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years,
* ACL-reconstructed using hamstring tendon auto-grafts, and a pathological defined between limb asymmetry ratio (operated/non-operated) of more than 10 % for maximal isometric strength of the knee flexors, at 1 year follow-up.

Exclusion Criteria:

* Other known pathology conditions in hip, knee, or ankle,
* BMI above 35, and
* Not understanding written Danish language.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in isometric maximal knee flexor muscle strength | 12 weeks (intervention period)
  Change, pre- and post intervention using stabilized maximal isometric dynamometry (in Nm)

SECONDARY OUTCOMES:
Change in isometric knee extensor strength | 12 weeks (intervention period)
  Change, pre- and post intervention using stabilized maximal isometric dynamometry (in Nm)
Change in isometric maximal hamstring to quadriceps strength ratio | 12 weeks (intervention period)
  Change, pre- and post intervention using stabilized maximal isometric dynamometry (in percentage)
Change in Self-perceived knee related function | 12 weeks (intervention period)
  Change, pre- and post intervention, using Patient reported outcomes (PROM) questionnaires (KOOS, Knee injury and Osteoarthritis Outcome Score, all subscales)

OTHER OUTCOMES:
Gait analysis | 12 weeks (intervention period)
  Change, pre- and post intervention (12 weeks) using 3-dimensional Vicon motion analysis
Counter movement jump | 12 week intervention period
  Change, pre- and post intervention (12 weeks) using 3-dimensional Vicon motion analysis (force Development)
Change in One-leg jump for distance | 12 week intervention period
  Change, pre- and post intervention (12 weeks) in jumping distance (in cm). Simple functional test.
Change in Quadriceps and hamstring morphologies | 12 week intervention period
  Change, pre- and post intervention (12 weeks) concerning volume, peak cross sectional area and length of muscle and tendon, using Magnetic resonance imaging (MRI)
Change in Rate of force Development (RFD) in maximal quadriceps and hamstring strenght | 12 week intervention period
  Change, pre- and post intervention (12 weeks) using maximal isometric dynamometry (Nm/millisecond)
Change in Self-perceived knee related function and symptoms | 12 week intervention period
  Change, pre- and post intervention (12 weeks) using Patient reported outcomes (PROM) questionnaires (IKDC, subjective knee evaluation form)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Holsgaard-Larsen, ass.proff, Study Director — Orthopaedic Research Unit, Institute of Clinical Research, SDU
Locations (1):
- Orthopaedic Research Unit, Institute of Clinical Research, SDU, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bregenhof B, Jorgensen U, Aagaard P, Nissen N, Creaby MW, Thorlund JB, Jensen C, Torfing T, Holsgaard-Larsen A. The effect of targeted exercise on knee-muscle function in patients with persistent hamstring deficiency following ACL reconstruction - study protocol for a randomized controlled trial. Trials. 2018 Jan 26;19(1):75. doi: 10.1186/s13063-018-2448-3. PMID 29373984

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02939677/SAP_001.pdf